CLINICAL TRIAL: NCT03615313
Title: A Clinical Study of PD-1 Antibody Expressing mesoCAR-T Cells for Patients With Mesothelin Positive Advanced Solid Tumors
Brief Title: PD-1 Antibody Expressing mesoCAR-T Cells for Mesothelin Positive Advanced Solid Tumor
Acronym: PAEMCMPAST
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cell Therapy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSY-IEC-4.0/18-09/02
Record Dates: First submitted 2018-06-28; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Advanced Solid Tumor
Keywords: mesothelin, PD-1, CAR T cells, solid tumor
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody expressing mesoCAR-T cells (Experimental): Patients will receive two cycles of PD-1 antibody expressing mesoCAR-T cells treatment. Every cycle, peripheral blood mononuclear cells (PBMC) are collected on day -18, CAR-T cells are cultured in a GMP standard workshop. Patients are given a three-day regimen of chemotherapy consisting of fludarabine and cyclophosphamide aimed to deplete the lymphocytes before cells infusion. Then the patients will receive an i.v.gtt infusion of PD-1 antibody expressing mesoCAR-T cells from day 1 to day 3 (±3days).
  Interventions: Biological: PD-1 antibody expressing mesoCAR-T cells

INTERVENTIONS:
Biological: PD-1 antibody expressing mesoCAR-T cells — Patients with mesothelin positive cancer will be infused the PD-1 antibody expressing mesoCAR-T cells. The modified mesoCAR-T cells can specifically kill mesothelin positive cancer cells and secrete PD-1 antibody, which could enhance the cytotoxicity of mesoCAR-T cells and activate the tumor infiltrating lymphocytes.

SUMMARY:
This is a single-arm, open-label, one center clinical study, to determine the safety and efficacy of infusion of autologous T cells engineered to target mesothelin and express PD-1 antibodies in adult patients with advanced recurrent or refractory malignant solid tumors, which were positive expression of mesothelin.

DETAILED DESCRIPTION:
This study will be conducted using a phase I/II trial design to assess the safety and efficacy of the PD-1 antibody expressing mesoCAR-T for patients with mesothelin positive, advanced recurrent or refractory malignant solid tumors. MesoCAR-T can specifically and effectively kill the mesothelin positive cancer cells, PD-1 antibody are secreted from the CAR-T cells could improve immunosuppression microenvironment, new CAR-T cells contain the advantages of CAR-T and immune checkpoint inhibitor, which is a promising therapeutic method for advanced solid tumors.

The new CAR-T therapy is applied to clinical practice as bellow. T cells are prepared from peripheral blood mononuclear cells (PBMC) by leukapheresis, and then activated and engineered to express chimeric antigen receptors (CARs) targeting mesothelin and PD-1 antibody. Cells are proliferated in culture and returned to the patients by venous transfusion therapy. A total of 50 patients may be enrolled in the study. The total duration of the study is expected to be approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory advanced solid malignancies (diagnosed by histology or cytology detection), including malignant mesothelioma, pancreatic cancer, bile duct cancer, ovarian cancer, lung cancer, gastric cancer, etc.
2. Patients who failed after second-line treatment, or who are unwilling to receive second-line treatment after failed to recieve first-line treatment.
3. Gender unlimited, age from 18 years to 80 years.
4. Life expectancy ≥ 3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Adequate venous access for Peripheral blood mononuclear cell (PBMC) apheresis, and no other contraindications.
7. Immunohistochemistry (IHC) score of mesothelin on tumor tissue ≥ 1+.
8. The requirements of laboratory examination: Neutrophilic granulocyte ≥ 1.0×10^9/L; Platelet ≥ 50×10^9/L; Hemoglobin ≥ 90g/L; total bilirubin ≤ 2 times the upper limit of the normal value; Alanine aminotransferase and Aspartate transaminase (ALT and AST) ≤ 2.5 times the upperlimit of the normal value (If there is liver metastasis, they should be ≤ 5 times the upperlimit of the normal value); Serum creatinine ≤ 1.5 times the upper limit of the normalvalue.
9. There is at least one measurable tumor lesion; According to RECIST 1.1 standard, it is suitable to evaluate the therapeutic response and progress of tumor.
10. Patients have adequate ability to understand, sign informed consents and take part in the clinical research voluntarily.
11. Female patients in child bearing period must have evidence of negative pregnancy test or male patients, and they agree to take effective contraceptive measures until 30 days after cells infusion.

Exclusion Criteria:

1. Patients with active viral or bacterial infection, and have failed to be controlled by anti-infective treatment.
2. Patients with seropositive response of Human immunodeficiency virus (HIV) and syphilis, or fail to control the hepatitis B virus or hepatitis C virus infection.
3. Patients who are undergoing treatment of autoimmune or organ transplantation diseases, or patients who need long-term use of immunosuppressive drugs such as glucocorticoid.
4. Patients with severe heart and lung dysfunction, high blood pressure and cannot be controlled with medicine, unstable coronary artery disease (uncontrolled arrhythmias, unstable angina pectoris), uncompensated congestive heart failure, myocardial infarction within six months.
5. Patients with any other illness that the investigators consider it will may affect the patient's treatments, follow-up or assessment, including any uncontrolled clinically significant neurological or psychiatric disorders, immunoregulatory diseases, metabolic diseases, infectious diseases and so on.
6. Received cancer treatment prior to enroll the group within the following time (including drug clinical trials):

(1) The withdrawal time of chemotherapy before enrollment was shorter than the treatment cycle of chemotherapy.

(2) The use of anti-tumor therapy within 4 weeks before the study or less than 5 times of the half-life period of the drugs (including radiation therapy, chemotherapy, small molecules and biological therapy or immunotherapy), the shortest period of time was as the criterion (but the shortest time should not be less than 21 days).

7. Women patients in pregnancy period or suckling period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-06 (Estimated); Primary Completion 2020-08-03 (Estimated); Study Completion 2020-12-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events of infusion of autologous PD-1 antibody expressing mesothelin-targeted CAR-Tcells | 2 years
  Incidence of treatment-related adverse events are assessed using the NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Objective response rate (ORR) of the treatment using PD-1 antibody expressing mesoCAR-T cells for advanced solid tumors | 2 years
  Objective response rate (ORR) of the treatment is assessed according to the response evaluation criteria in solid tumor version 1.1 (RECIST1.1), which contains complete response (CR) and partial response (PR).
Progression free survival | 2 years
  Progression free survival is defined as the time from the day in which the patient is enrolled to the date on which tumor progresses or the date on which the patient dies for any cause.
Overall survival | 2 years
  Overall survival is defined as the time from the day in which the patient is enrolled to the date on which the patient dies for any cause.

OTHER OUTCOMES:
Proliferation and persistence of mesothelin specific CAR-T cells in peripheral blood of the patients | 6 months
  CAR-T proportionin in peripheral blood of the patients is detected by flow cytometry assay to study the proliferation and persistence of mesothelin specific CAR-T cells.
PD-1 antibody level in peripheral blood of the patients after treatment | 6 months
  PD-1 antibody level are detected by ELISA assay to assess the expressing level of PD-1 antibody from CAR-T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Qian, PhD, Study Chair — Shanghai Cell Therapy Research Institute; Huajun Jin, PhD, Study Chair — Shanghai Cell Therapy Research Institute; Qing Xu, PhD, Principal Investigator — Shanghai 10th People's Hospital; Zhiwei Zhang, PhD, Study Director — Shanghai Cell Therapy Research Institute; Yan Sun, Study Director — Shanghai Cell Therapy Research Institute; Huimei Li, PhD, Study Director — Shanghai Cell Therapy Research Institute; Juemin Fang, PhD, Principal Investigator — Shanghai 10th People's Hospital; Song Gao, PhD, Principal Investigator — Shanghai 10th People's Hospital; Xianling Guo, Principal Investigator — Shanghai 10th People's Hospital; Hui Wang, Principal Investigator — Shanghai 10th People's Hospital; Zhongzheng Zhu, Principal Investigator — Shanghai 10th People's Hospital; Jianhua Chen, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- China, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fang J, Ding N, Guo X, Sun Y, Zhang Z, Xie B, Li Z, Wang H, Mao W, Lin Z, Qin F, Yuan M, Chu W, Qin H, Qian Q, Xu Q. alphaPD-1-mesoCAR-T cells partially inhibit the growth of advanced/refractory ovarian cancer in a patient along with daily apatinib. J Immunother Cancer. 2021 Feb;9(2):e001162. doi: 10.1136/jitc-2020-001162. PMID 33589520